CLINICAL TRIAL: NCT05300308
Title: Lymphoedema and Nocturia/ Nocturnal Polyuria After Pelvic Lymph Node Dissection (LND): Prospective Observational Study
Brief Title: Lymphoedema and Nocturia/Nocturnal Polyuria After Pelvic LND for Urogenital Cancer
Acronym: UroLymph
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s66072
Record Dates: First submitted 2022-01-17; First posted 2022-03-29 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Urogenital Cancer; Lower Limb Lymphedema; Nocturia; Nocturnal Polyuria
MeSH Terms: conditions — Urogenital Neoplasms; Nocturia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- transperitoneal pelvic lymph node dissection for treatment of urogenital cancer: patients planned for transperitoneal pelvic lymph node dissection for treatment of urogenital cancer (including prostate or bladder cancer)
  Interventions: Other: usual care

INTERVENTIONS:
Other: usual care — The information about lymphoedema and its prevention is given during the hospital stay by the physical therapist of the department of urology. Skincare consists of daily skin moisturizer of feet and legs and prevention and care of wounds. Active exercises are performed to gain endurance and muscle strength after surgery and to stimulate the blood and lymph circulation. The exercises are supervised by the home physical therapist. Frequency of the supervised exercises is gradually decreased. If a patient develops lymphoedema, he/she receives compression stockings.

SUMMARY:
After the treatment of urogenital cancer, a person may develop lymphoedema of the leg(s) and/ or midline region. Clinical symptoms include abnormal tissue swelling, sensation of limb heaviness, erythema, pain, and impaired limb function. Lymphoedema can have a negative impact on quality of life (QoL) and the impact of lymphoedema on the cancer treatment decision making process is underestimated. A limited number of studies have evaluated the incidence rate of midline and leg lymphoedema after surgery for urogenital cancers and have investigated the prognostic variables. In addition, to the researchers knowledge, no evidence exists regarding which (combination of) clinical measuring methods are most sensitive to detect early lymphoedema at the lower limbs after the treatment of urogenital cancer. Therefore, in this prospective observational study, the epidemiology (i.e. incidence/ prevalence rate and prognostic variables) and the detection methods of lower limb lymphoedema after pelvic lymph node dissection for urogenital cancer will be investigated.

Additionally, the epidemiology of nocturia and nocturnal polyuria will be studied (since this information is also missing in literature).

DETAILED DESCRIPTION:
Lymphoedema is caused by malfunction of the lymphatic system whether or not in combination with extra load on this system. Some patients develop lymphoedema after treatment for cancer: secondary lymphoedema or acquired lymphoedema. In 2018, 11 645 patients in Belgium were diagnosed with urogenital cancer cancer, including prostate and bladder cancer. A possible treatment consists of prostatectomy or cystectomy in combination with transperitoneal pelvic lymph node dissection. Patients who undergo treatment for cancer may develop lower limb lymphoedema or lymphoedema at midline. To the researchers knowledge, investigation of incidence of lower limb lymphoedema (LLL) is limited. Also, the prognostic variables for the development of LLL are unknown. Furthermore, no scientific evidence consists regarding which (combination of) clinical measurement methods are most sensitive to detect early LLL after transperitoneal pelvic lymph node dissection. Thresholds to identify subclinical lymphoedema in one or both legs are lacking. Besides lymphoedema in the lower limbs, treatment for cancer also often results in urinary problems. Especially urinary stress incontinence has been described in literature. However, in clinical practice, it is clear that prostatectomy is often associated with other urinary complications, as nocturia and nocturnal polyuria. To the researchers knowledge, there are no trials investigating the prognostic variables for the development of nocturia/ nocturnal polyuria after transperitoneal pelvic lymph node dissection for urogenital cancer.

Therefore, the researchers will execute a trial investigating the epidemiology (i. e incidence, prevalence and prognostic variables), detection methods and the feasibility of a trial about the early treatment of LLL after transperitoneal pelvic lymph node dissection for urogenital cancer. The epidemiology of LLL, nocturia and nocturnal polyuria will be investigated.

Participants: 150 patients undergoing a transperitoneal pelvic lymph node dissection for urogenital cancer will be included. These participants will be followed-up from baseline (pre-surgery) until 1 year post-surgery. All participants are evaluated at the University Hospitals Leuven, campus Gasthuisberg.

Procedure: The potential participant will be screened first to see if the patients meets the inclusion criteria. After signing the informed consent form, the participant will be followed in the prospective observational trial. The duration of the prospective observational trial is 2 years. Participants can be included until 1 year after the start of the trial.

Evaluation: There will be clinical evaluation of lymphoedema as well as treatment for lymphoedema. Participants in the prospective observational trial will be evaluated 4 times: baseline (pre-surgery), 6 weeks, 6 and 12 months post-surgery.

Treatment: All participants in the prospective observational trial receive standard of care. This consists out of information, skincare and exercises. The information about lymphoedema and its prevention is given by the physical therapist of the department of urology during the hospital stay. Skincare consists of daily moisturizer of legs and feet and prevention and care of wounds. The exercises are supervised by the home physical therapist. The frequency of the session at the physical therapist are gradually decreased.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic urogenital cancer (i.e. prostate cancer or bladder cancer)
* Planned transperitoneal pelvic lymph node dissection or salvage lymph node dissection
* Salvage lymph node dissection
* Before inclusion, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Radiological evidence of metastatic disease based on pelvic CT/MRI and bone scan
* Clinical signs of chronic venous insufficiency (CEAP C3-C6)
* History of lymph node dissection/ radiotherapy at the level of the pelvis or groin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients planned for transperitoneal pelvic lymph node dissection for treatment of urogenital cancer (including prostate or bladder cancer)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence rate of lower limb lymphoedema after urogenital cancer (i.e. number of patients with newly diagnosed lower limb lymphoedema) 6 weeks post-surgery | 6 weeks post-surgery
  Calculation of the proportion of patients who developed leg lymphoedema during a certain time interval (defined as 5.0% or more increase of the leg volume) and calculation of the proportion of patients who developed midline lymphoedema during a certain time interval (defined as 20% or more increase of the baseline water content at the prepubic region)
Cumulative incidence rate of lower limb lymphoedema after urogenital cancer (i.e. number of patients with newly diagnosed lower limb lymphoedema) 6 months post-surgery | 6 months post-surgery
  Calculation of the proportion of patients who developed leg lymphoedema during a certain time interval (defined as 5.0% or more increase of the leg volume) and calculation of the proportion of patients who developed midline lymphoedema during a certain time interval (defined as 20% or more increase of the baseline water content at the prepubic region)
Cumulative incidence rate of lower limb lymphoedema after urogenital cancer (i.e. number of patients with newly diagnosed lower limb lymphoedema) 12 months post-surgery | 12 months post-surgery
  Calculation of the proportion of patients who developed leg lymphoedema during a certain time interval (defined as 5.0% or more increase of the leg volume) and calculation of the proportion of patients who developed midline lymphoedema during a certain time interval (defined as 20% or more increase of the baseline water content at the prepubic region)
Prognostic value of 'baseline age' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Dependent variable = presence of leg lymphoedema/ presence of midline lymphoedema Independent variable= Age (years) will be self-reported through interview.
Prognostic value of ' Baseline fat mass' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Baseline fat mass will be measured using Bio-impedance Spectroscopy
Prognostic value of ' Baseline physical activity level' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Baseline physical activity level will be assessed with the International Physical Activity Questionnaire (IPAQ).
  The IPAQ is a 27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Prognostic value of ' Baseline educational level' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Educational level will be self-reported through interview.
Prognostic value of ' baseline comorbidities' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Comorbidities will be reported through a self-developed co-morbidity questionnaire, based on IDEWE questionnaire.
Prognostic value of 'type of cancer' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Information regarding the type of urogenital cancer (prostate versus bladder) and the stage of the urogenital cancer is collected (i.e. histological subtype, PSA (if PCa), pTN stage, ISUP grade group (if PA); by exploring the patient's medical file.
Prognostic value of 'Tumor stage' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Information regarding the type of urogenital cancer (prostate versus bladder) and the stage of the urogenital cancer is collected (i.e. histological subtype, PSA (if PCa), pTN stage, ISUP grade group (if PA); by exploring the patient's medical file.
Prognostic value of 'Lymph node stage' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Information regarding the type of urogenital cancer (prostate versus bladder) and the stage of the urogenital cancer is collected (i.e. histological subtype, PSA (if PCa), pTN stage, ISUP grade group (if PA); by exploring the patient's medical file.
Prognostic value of 'number of positive lymph nodes' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Number of positive lymph nodes is collected through the patient's medical file.
Prognostic value of 'postoperative complications' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Information regarding the complications related to the surgery as well as adjuvant therapies is collected. Surgical complications will be assessed according to the Clavien-Dindo Classification of Surgical Complications.
Prognostic value of 'type of lymph node dissection' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Cancer treatment characteristics are collected (i.e. type of surgery, type of lymph node dissection, number of lymph nodes removed, presence of postoperative drain, number of positive lymph nodes, adjuvant therapies; by exploring the patient's medical file.
  Type of lymph node dissection: Limited- Standard- Extended- Super extended
Prognostic value of 'number of lymph nodes removed' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Cancer treatment characteristics are collected (i.e. type of surgery, type of lymph node dissection, number of lymph nodes removed, presence of postoperative drain, number of positive lymph nodes, adjuvant therapies; by exploring the patient's medical file.
Prognostic value of 'Adjuvant Radiotherapy' for the development of lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Cancer treatment characteristics , including adjuvant radiotherapy are collected; by exploring the patient's medical file.

SECONDARY OUTCOMES:
Point prevalence rate of lower limb lymphoedema (i.e. number of patients with lower limb lymphoedema) | up to 12 months post-surgery
  Calculation of the proportion of patients with leg lymphoedema at a certain time point (defined as 5.0% or more increase of the leg volume) and calculation of the proportion of patients with midline lymphoedema at a certain time point (defined as 20% or more increase of the baseline water content at the prepubic region): 6 weeks, 6 and 12 months post-surgery
Reliability of detection lower limb lymphoedema developing after the treatment of urogenital cancer | 12 months post-surgery
  To investigate reliability, all participants with lower limb lymphoedema at 12 months post-surgery will be evaluated three times with each evaluation method: intra and interrater reliability will be determined
Time efficiency of lymphoedema measurements | 12 months post-surgery
  To determine feasibility of each method, time efficiency will be examined for each method: setup time (time needed to prepare the measurement), execution time ( time needed for a bilaterally execution of the measurement) and total time (required for the setup and the execution of the measurement) (min, sec)
Presence of limitations of lymphoedema measurements | 12 months post-surgery
  limitations regarding clinical feasibility will be listed and scored (yes/no) for each method.
Validity of lymphoedema measurements | 12 months post-surgery
  As "gold standard" to compare the different measurement methods with, every patient will be evaluated individually once by the project's international expert panel, during a monthly (virtual) meeting (2 up to 3h). They will decide whether patients should be labelled as showing 'presence of early signs of lower limb lymphoedema (1)' or 'no signs (0)'. Decision making will occur with an initial assessment of the experts, i.e. in advance of the monthly meeting. Then the project manager will lead the meeting on the basis of the assessments and subsequently conduct a new 'vote'. In case >2/3 of the experts (= clear majority) decides a patient should receive a diagnosis of lymphoedema, then this patient receives the diagnosis.
diagnostic accuracy of the screening methods for lower limb lymphoedema | 12 months post-surgery
  outcomes resulting from the measurement method will be compared against the yes/no score regarding clinical presence of LLL from our international expert group
Point prevalence rate of nocturia and nocturnal polyuria | up to 12 months post-surgery
  Calculation of the proportion of patients with nocturia/ nocturnal polyuria at a certain time point: baseline, at 6 weeks, 6 and 12 months post-surgery
Prognostic value of 'baseline age' for the development of nocturia and nocturnal polyuria | 12 months
  Age (years) will be self-reported through interview
Prognostic value of 'late-night fluid intake' for the development of nocturia and nocturnal polyuria | 12 months
  late-night fluid intake will be assessed through the micturition chart that (during 24 hours, in the week prior to the assessment visit) has to be filled in by the patient before surgery and at 6 weeks, 6 months and 12 months after surgery. The patient has to write down the time, frequency and quantity of urinating during the day and night. The time of drinking a consumption, the amount of a consumption and which consumption also has to be recorded.
Prognostic value of 'late-night caffeine/alcohol use (3 hours before going to bed)' for the development of nocturia and nocturnal polyuria | 12 months
  late-night caffeine/alcohol use (3 hours before going to bed) will be assessed through the micturition chart that (during 24 hours, in the week prior to the assessment visit) has to be filled in by the patient before surgery and at 6 weeks, 6 months and 12 months after surgery. The patient has to write down the time, frequency and quantity of urinating during the day and night. The time of drinking a consumption, the amount of a consumption and which consumption also has to be recorded.
Prognostic value of 'comorbidities' for the development of nocturia and nocturnal polyuria | 12 months
  Comorbidities will be reported through a self-developed co-morbidity questionnaire, based on IDEWE questionnaire.
Prognostic value of 'baseline fat mass' for the development of nocturia and nocturnal polyuria | 12 months
  Baseline fat mass will be measured using Bio-impedance Spectroscopy
Prognostic value of 'baseline physical activity' for the development of nocturia and nocturnal polyuria | 12 months
  Baseline physical activity level will be assessed with the International Physical Activity Questionnaire (IPAQ).
  The IPAQ is a 27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old.
Prognostic value of 'baseline educational level' for the development of nocturia and nocturnal polyuria | 12 months
  Educational level will be self-reported through interview.
Prognostic value of 'type of cancer' for the development of nocturia and nocturnal polyuria | 12 months
  information regarding the type of urogenital cancer (prostate versus bladder) and the stage of the urogenital cancer is collected (i.e. histological subtype, PSA (if PCa), pTN stage, ISUP grade group (if PA); by exploring the patient's medical file.
Prognostic value of 'tumor stage' for the development of nocturia and nocturnal polyuria | 12 months
  information regarding the type of urogenital cancer (prostate versus bladder) and the stage of the urogenital cancer is collected (i.e. histological subtype, PSA (if PCa), pTN stage, ISUP grade group (if PA); by exploring the patient's medical file.
Prognostic value of 'lymph node stage' for the development of nocturia and nocturnal polyuria | 12 months
  information regarding the lymph node stage is collected by exploring the patient's medical file.
Prognostic value of 'number of positive lymph nodes' for the development of nocturia and nocturnal polyuria | 12 months
  Number of positive lymph nodes is collected through the patient's medical file.
Prognostic value of 'postoperative complications' for the development of nocturia and nocturnal polyuria | 12 months
  Surgical complications will be assessed according to the Clavien-Dindo Classification of Surgical Complications. Complications will be determined as 30-day, 90-day or late (>90 days) complications.
Prognostic value of 'type of lymph node dissection' for the development of nocturia and nocturnal polyuria | 12 months
  Information about the type of lymph node dissection is collected by exploring the patient's medical file.
  Type of lymph node dissection: Limited- Standard- Extended- Super extended
Prognostic value of 'number of lymph nodes removed' for the development of nocturia and nocturnal polyuria | 12 months
  number of lymph nodes removed: by exploring the patient's medical file.
Prognostic value of 'radiotherapy' for the development of nocturia and nocturnal polyuria | 12 months
  Cancer treatment characteristics , including radiotherapy are collected; by exploring the patient's medical file.
Prognostic value of 'presence of postoperative drain' for the development of nocturia and nocturnal polyuria | 12 months
  Cancer treatment characteristics are collected, including the presence of postoperative drain, are collected by exploring the patient's medical file.
Prognostic value of 'presence of lymphoedema' for the development of nocturia and nocturnal polyuria | 12 months
  The presence of leg lymphoedema (defined as 5.0% or more increase of the leg volume) and midline lymphoedema (defined as 20% or more increase of the baseline water content at the prepubic region)

CONTACTS AND LOCATIONS:
Overall Officials: Nele Devoogdt, Prof. Dr., Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, campus Gasthuisberg, Leuven, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided